CLINICAL TRIAL: NCT00002301
Title: Foscarnet Treatment of Cytomegalovirus (CMV) Retinitis in AIDS Patients Not Eligible for Ganciclovir Therapy and Ganciclovir Treatment Failures
Brief Title: A Study of Foscarnet in the Treatment of Cytomegalovirus (CMV) of the Eyes in Patients With AIDS Who Have Not Had Success With Ganciclovir
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Astra USA (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 020B; 88-FOS-02
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1991-03

CONDITIONS: Cytomegalovirus Retinitis; HIV Infections
Keywords: Retinitis; AIDS-Related Opportunistic Infections; Ganciclovir; Foscarnet; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome; Antiviral Agents
MeSH Terms: conditions — Cytomegalovirus Retinitis; HIV Infections; Retinitis; AIDS-Related Opportunistic Infections; Multiple Acyl Coenzyme A Dehydrogenase Deficiency; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome | interventions — Foscarnet

INTERVENTIONS:
Drug: Foscarnet sodium

SUMMARY:
To evaluate the safety and efficacy of foscarnet induction treatment of cytomegalovirus (CMV) retinitis in AIDS patients who have previously suffered severe dose-limiting ganciclovir-related myelosuppression, who are ineligible for ganciclovir treatment due to myelosuppression or who have clearly failed to have a therapeutic response to ganciclovir therapy. To assess the duration of clinical response. To evaluate the effect on quantitative CMV cultures of blood and urine. To determine the effect on recovery of HIV p24 antigen capture direct from plasma.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Ganciclovir.

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Known allergy to foscarnet.
* Any clinically significant pulmonary or neurologic impairment (e.g., patients who are intubated or comatose).
* Corneal, lens, or vitreous opacification which precludes examination of the fundi in patients with cytomegalovirus (CMV) retinitis.

Concurrent Medication:

Excluded:

* Acyclovir.
* Nephrotoxic agent.

Patients with the following are excluded:

* Known allergy to foscarnet.
* Any clinically significant pulmonary or neurologic impairment (e.g., patients who are intubated or comatose).
* Corneal, lens, or vitreous opacification which precludes examination of the fundi in patients with CMV retinitis.

Prior Medication:

Excluded within 7 days of study entry:

* Immunomodulators.
* Biologic response modifiers.
* Investigational agents.

AIDS patients experiencing cytomegalovirus (CMV) retinitis may be enrolled if they meet one of the following criteria:

* Myelosuppression:
* Previously suffered severe dose-limiting ganciclovir-related myelosuppression, or are ineligible for ganciclovir treatment due to myelosuppression.
* Ganciclovir treatment failure:
* Clearly failed to have a therapeutic response to ganciclovir therapy.
* Patients must be able to give informed consent.
* Patients presenting with a baseline absolute neutrophil count < 750 cells/mm3 or baseline platelet count < 50000 platelets/mm3 will be categorized as ineligible to receive ganciclovir induction therapy and will be allowed to enter the study.
* Patients who enter the study because of ganciclovir toxicity will have received ganciclovir therapy which resulted in either absolute neutrophil count falling to < 750 cells/mm3 or platelet count falling to < 50000 platelets/mm3 on two separate occasions during either

  1) a ganciclovir induction regimen of 7.5 mg or less ganciclovir/kg/day in divided doses or 2) a maintenance regimen of 5 mg or less ganciclovir/kg/day as a single dose.
* Patients who enter the study because of ganciclovir treatment failure will meet one of the following criteria:
* 1) CMV retinitis progression as defined in section V.C.1., i.e., has occurred either at the end of a 10 - 21 day induction course of ganciclovir (7.5 - 10.0 mg/kg/day in divided doses) or 2) during the first 28 days of maintenance ganciclovir therapy (5 or more mg/kg/day in at least 5 days/week) where maintenance therapy began within

  1. week of completing induction therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Foscarnet Research Program / Park Plaza Hosp, Houston, Texas, United States

REFERENCES:
- [Background] Ussery FM, Karol C, Conklin R, Gathe J, Stool E, Redding K. Preliminary results from an on-going prospective evaluation of foscarnet in the treatment of AIDS-associated cytomegalovirus retinitis. Int Conf AIDS. 1989 Jun 4-9;5:551 (abstract no MCP60)